CLINICAL TRIAL: NCT04731532
Title: University of Health Sciences Bursa Yuksek Ihtisas Education and Training Hospital
Brief Title: Comparison of Thoracic Vibration With Classical Respiratory Physiotherapy in Patients With Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Seyhan Dülger,MD, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2018/04-02
Record Dates: First submitted 2018-06-20; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Medicine; Ventilators, Mechanical
Keywords: respiratory physiotherapy

STUDY DESIGN:
Intervention Model Description: randomized, controlled study
Who Masked: Participant, Care Provider
Masking Description: pulmonary department, physical therapy and rehabilitation, anesthesiology and reanimation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical respiratory physiotherapy application (Active Comparator): Patient positions, postural drainage application tapping and trifled
  Interventions: Procedure: classical respiratory physiotherapy with thoracic vibration
- classical respiratory physiotherapy with thoracic vibration (Active Comparator): Thoracic Vibration: The physiotherapist places his hands open with his / her fingers on the front and side walls of the patient's chest when the elbow is at 5-10 degrees of flexion. The elbow expands the patient's chest with vibrations. Exercise can be repeated 5-10 times a day+Patient positions, postural drainage application tapping and trifled
  Interventions: Procedure: classical respiratory physiotherapy with thoracic vibration

INTERVENTIONS:
Procedure: classical respiratory physiotherapy with thoracic vibration — Classical respiratory physiotherapy application: Patient is positioned, postural drainage application is operated by tapping and trifled .
  Other Names: classical respiratory physiotherapy

SUMMARY:
Inclusion and Exclusion Criteria: Patients aged 18-65 years who are admitted to the investigator's 3rd Stage Intensive Care Unit and are dependent on mechanical ventilation will be included. The study was planned with 80 patients. Those with known chronic illnesses such as renal insufficiency, heart failure, liver failure, diabetes mellitus, hypertension, chronic obstructive pulmonary disease etc.,; patients in intensive care for postoperative follow-up; patients with mechanical ventilation due to chest or abdominal trauma will be excluded from the study.

Patients who meet the study criteria will be evaluated by a physiotherapy and rehabilitation specialist and will be decided to be included in the respiratory physiotherapy program. The patients will be treated by two physiotherapists in the intensive care unit at random. One of the physiotherapists will perform classical respiratory physiotherapy with thoracic vibration and the other will only perform classical respiratory physiotherapy.

Patients' acute physiology and chronic health assessment II (APACHE II) scores, partial oxygen pressure(PaO2) /fraction of inspired oxygen inspired oxygen fraction (FiO2), tidal volume, minute respiratory rate, peak air pressure, mean air pressure, blood lactate levels will be recorded daily. These values will be collected in the daily routine of the illness depending on the mechanical ventilation, by recording the already performed operations to follow the patient's clinic. If the duration of the total mechanical ventilation and complications occur, the type and timing of the complications will be examined.

At the end of the study, both physiotherapy methods, APACHE II scores, PaO2 / FiO2 values, tidal volume required, minute respiratory rate, peak air pressure, mean air pressure, blood lactate levels, mechanical ventilation duration and complications will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* Patients who accepted for Step 3 Intensive Care Unit and connected to mechanical ventilation

Exclusion Criteria:

* Patients with known chronic disease;
* Patients in intensive care for postoperative follow-up;
* Patients with mechanical ventilation due to chest or abdominal trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-25 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Duration of patient waking from the mechanical ventilator | through study completion, an average of 1 year
  hour
Measuring of chronic health assessment II (APACHE II) scores | through study completion, an average of 1 year
  score
Determination of tidal volume | through study completion, an average of 1 year
  mmHg
Measuring of minute respiratory rate | through study completion, an average of 1 year
  counts / minute
Determination of peak air pressure | through study completion, an average of 1 year
  mmHg
Determination of mean air pressure | through study completion, an average of 1 year
  mmHg
Measuring of blood lactate levels | through study completion, an average of 1 year
  mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Seyhan Dülger, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://doi.org/10.1016/j.aucc.2017.10.001